CLINICAL TRIAL: NCT04739137
Title: Development and Validation of a Smart-tv Application for the Self Examination of the Distance Visual Acuity in Macular Edema Patients
Brief Title: Smart-TV Application for the Self Examination of the Distance Visual Acuity in Macular Edema Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES1/Th5/21-1-2021
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Low Vision; Macular Edema; Refractive Errors
Keywords: smart features; Smart-tv App
MeSH Terms: conditions — Vision, Low; Macular Edema; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 100 patients with diagnosed macular edema will be enrolled
  Interventions: Diagnostic Test: DDiVAT Testing; Diagnostic Test: Distance visual acuity assessment via ETDRS chart

INTERVENTIONS:
Diagnostic Test: DDiVAT Testing — Participants will self examine his/her distance visual acuity via application in a simulation room of our department with certain predetermined environmental lighting conditions using the same smart devices.
Diagnostic Test: Distance visual acuity assessment via ETDRS chart — The distance visual acuity of each participant will be measured with the conventional method via ETDRS chart

SUMMARY:
Primary objective of our study is the development and validation of an application for smart-TVs for the self-examination of the distant visual acuity of patients diagnosed with macular edema.

DETAILED DESCRIPTION:
Present study aims to develop and validate an application installed in Smart-TVs. This application will be referred to patients suffering from macular edema, allowing the self-examination of the patient in terms of distant visual acuity. The development of a simple but reliable way of self-examination of distant visual acuity would bring beneficial results in the overall management of these patients as significantly would reduce the flows to the outpatient ophthalmology clinics of the NSS Hospitals, would serve the purposes of the social distancing imposed by the current state of the pandemic but also any analogous situation and would help the patient to be vigilant and actively involved in the management of his disease.

ELIGIBILITY:
Inclusion Criteria:

* age-dependent macular degeneration
* diabetic macular edema

Exclusion Criteria:

* corneal diseases
* glaucoma
* psychiatric disorders
* inability to cooperate

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal- and low-sighted participants aged 40 to 85 years
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Distance visual acuity test via ETDRS chart | 1 week
  The distance visual acuity of each participant will be evaluated by the same examiner
Distance visual acuity self assessment via DDiVAT | 1 week
  Participants will self examine his/her distance visual acuity via application in a simulation room of our department with certain predetermined environmental lighting conditions using the same smart devices.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, Study Chair — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: Undecided